CLINICAL TRIAL: NCT02445378
Title: The Effect of Aromatherapy on Insomnia and Other Common Cancer Patient Symptoms
Brief Title: Aromatherapy and Essential Oils in Improving Insomnia and Other Symptoms in Patients With Newly Diagnosed Acute Leukemia Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Lisa Blackburn, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: OSU-14182; NCI-2015-00549 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Acute Leukemia; Anorexia; Anxiety; Depression; Dyspnea; Insomnia; Nausea; Pain
Keywords: Aromatherapy; essential oils; Acute Leukemia
MeSH Terms: conditions — Anorexia; Anxiety Disorders; Depression; Dyspnea; Sleep Initiation and Maintenance Disorders; Nausea; Pain | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (aromatherapy and essential oils week 1) (Experimental): Patients select between 3 scented essential oils: peppermint, lavender, or chamomile which is diffused in the hospital room from approximately 9 PM in the evening until morning during week 1 and placebo intervention using rose water during week 2.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Placebo; Other: Questionnaire Administration
- Group II (aromatherapy and essential oils week 3) (Experimental): Patients undergo placebo intervention using rose water during week 1 and aromatherapy and essential oils as in Group I during week 2.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Aromatherapy and Essential Oils — Undergo aromatherapy and essential oils
  Other Names: Aromatherapy
Other: Placebo — Undergo placebo intervention using rose water
  Other Names: placebo therapy; PLCB; sham therapy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies aromatherapy and essential oils in improving insomnia and other symptoms in patients with newly diagnosed acute leukemia. Aromatherapy and essential oils may help improve insomnia and other complications caused by chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Does the addition of aromatherapy by diffusion of essential oils improve insomnia in newly diagnosed, hospitalized leukemia patients?

SECONDARY OBJECTIVES:

I. Does the addition of aromatherapy by diffusion of essential oils improve other common symptoms in newly diagnosed, hospitalized leukemia patients, including pain, nausea, lack of appetite, shortness of breath, depression, anxiety and wellbeing? II. Do newly diagnosed, hospitalized leukemia patients find the use of aromatherapy for symptom management a positive experience?

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients select between 3 scented essential oils: peppermint, lavender, or chamomile which is diffused in the hospital room from approximately 9 PM in the evening until morning during week 1 and placebo intervention using rose water during week 2.

GROUP II: Patients undergo placebo intervention using rose water during week 1 and aromatherapy and essential oils as in Group I during week 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are newly diagnosed with acute leukemia and hospitalized to receive their initial 4 weeks of intensive induction chemotherapy for this disease

Exclusion Criteria:

* Asthma or other reactive airway disease
* Sleep apnea
* Planned less than two week hospitalization
* Change in pain medications/sleeping medications/anxiety medications/antiemetics during the trial
* Patients who have not completed their initial steroids
* Patients who are confused and unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12-28 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11-05 (Actual)

PRIMARY OUTCOMES:
Improvement of Insomnia graded by Pittsburgh Sleep Quality Index (PSQI) | 1 month
  Statistical analysis will be performed using a mixed effects linear regression model. This model is designed to test the effects of interest (i.e., the effect of aromatherapy relative to baseline and to placebo) while accounting for the within-subject correlation arising from the repeated measures design. A 20% positive change in PSQI score will be seen as significant.

SECONDARY OUTCOMES:
Improvement of common symptoms including pain, nausea, lack of appetite, shortness of breath, depression, anxiety, and wellbeing graded by Edmonton Symptom Assessment Scale - revised (ESASr) | Baseline to 2 weeks
Rate of positive experience with aromatherapy | Up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Blackburn, MS,RN,AOCNS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu